CLINICAL TRIAL: NCT07300748
Title: The Effectiveness of Cardiopulmonary Exercise in Children With Pectus Excavatum: A Single-Blind, Randomised Controlled Trial
Brief Title: Effectiveness of Cardiopulmonary Exercises for Children With Pectus Excavatum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Naz Kalem, PM&R Specialist, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-168
Record Dates: First submitted 2025-11-13; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pectus Excavatum Deformity
Keywords: pectus excavatum; cardiopulmonary exercises
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cardiopulmonary exercises group at hospital (Experimental): The working group will be provided with a personalised exercise plan by a physiotherapist specialising in that field at the cardiopulmonary rehabilitation unit, to be carried out twice a week for five weeks. Patients will work on a bicycle ergometer. In addition, the same physiotherapist will demonstrate breathing and posture exercises for patients to perform at home.
  Interventions: Other: Cardiopulmonary exercises at hospital
- pulmonary exercises group at home (Active Comparator): The physiotherapist will only demonstrate the breathing and posture exercises that patients in the control group will perform at home.
  Interventions: Other: Pulmonary and posture exercises at home

INTERVENTIONS:
Other: Cardiopulmonary exercises at hospital — Patients will exercise using a bicycle ergometer. In addition, the same physiotherapist will demonstrate breathing and posture exercises for them to perform at home.
  Arms: cardiopulmonary exercises group at hospital
Other: Pulmonary and posture exercises at home — The physiotherapist will demonstrate the breathing and posture exercises to be performed at home.
  Arms: pulmonary exercises group at home

SUMMARY:
The aim of this study is to investigate the effects of cardiopulmonary rehabilitation on respiratory function, exercise tolerance and posture in patients with pectus excavatum.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 5-18 years with pectus excavatum deformity
2. Children undergoing conservative treatment (vacuum orthosis, exercise)
3. Patients whose families have signed a consent form agreeing to participate in the study

Exclusion Criteria:

1. Known cardiac disease
2. Presence of an additional syndrome (Marfan syndrome, etc.)
3. Cobb angle ≥10°
4. Refusal to participate in the study
5. Presence of mixed deformity (pectus arcuatum)
6. Those with an indication for surgery

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiration and expiration pressure | first day of exercises program and 5th week of exercises program

SECONDARY OUTCOMES:
6 minute walking test | first day of exercises program and 5th week of exercises program
New York Posture Scale | first day of exercises program and 5th week of exercises program
Measurement of chest expansion in centimetres using a tape measure | first day of exercises program and 5th week of exercises program
Assessment of symptoms (exercise intolerance, psychological impact, resting dyspnoea, chest pain, spinal pain, gastrointestinal symptoms, palpitations, dyspnoea) using a visual analogue scale | first day of exercises program and 5th week of exercises program
Cobb angle analysis using the Diers Formatrix 4D device (Wiesbaden, Germany) | first day of exercises program and 5th week of exercises program
Thoracic kyphosis angle | first day of exercises program and 5th week of exercises program
body lenght | first day of exercises program and 5th week of exercises program
Saggital balance angle using the Diers Formatrix 4D device (Wiesbaden, Germany) | first day of exercises program and 5th week of exercises program
Coronal balance angle using the Diers Formatrix 4D device (Wiesbaden, Germany) | first day of exercises program and 5th week of exercises program
pelvic obliquity angle using the Diers Formatrix 4D device (Wiesbaden, Germany) | first day of exercises program and 5th week of exercises program

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)